CLINICAL TRIAL: NCT01830153
Title: A Phase II Multicenter Trial of RAD001 in Patients With Metastatic or Recurrent Sarcomas
Brief Title: RAD001 in Advanced Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Jin-Hee Ahn, Professor, Asan Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001CKR13T
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Last update posted 2013-04-12 (Estimated); Status verified 2013-04

CONDITIONS: Soft Tissue Sarcomas; Bone Sarcomas
Keywords: Soft tissue sarcomas; Bone sarcomas; RAD001; Refractory to conventional chemotherapy
MeSH Terms: conditions — Sarcoma; Bone Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 (Experimental): RAD001 was given as 10 mg orally once daily, and one cycle was defined as 28 days.
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001
  Other Names: Everolimus

SUMMARY:
This trial intends to test the efficacy and safety of RAD001 in patients with advanced sarcoma who failed to conventional chemotherapy.

DETAILED DESCRIPTION:
This multicenter, phase II trial evaluated the efficacy and safety of everolimus in patients with metastatic or recurrent bone and soft tissue sarcoma after failure of anthracycline and/or ifosfamide.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed metastatic, unresectable bone or soft tissue sarcomas who had past treatment with anthracycline and/or ifosfamide to which the disease was primarily refractory or progressed after initial response.
* Any of above drugs is allowed to be used as adjuvant treatment.
* Unidimensionally measurable disease
* 3 or less than prior chemotherapies
* Age 17 years old or older
* ECOG performance status 2 or less, Life expectancy 6 month or less
* Adequate bone marrow, liver, kidney, and cardiac function
* Written informed consent

Exclusion Criteria:

* Pregnant or lactating patients
* Patients with resectable metastasis
* Patients with history of CNS metastasis
* Gastrointestinal stromal tumors, chondrosarcoma, neuroblastoma
* Hypersensitivity to the active substance, to other rapamycin derivatives, or to any of the excipients.
* Any preexisting medical condition of sufficient severity to prevent full compliance with the study

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2010-04; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival rate at 16 weeks | 16 weeks
  Determined as the proportion of progression-free (complete response, partial response and stable disease) at 16 weeks of treatment

SECONDARY OUTCOMES:
Progression-free survival | Up to 24 months
  Defined as the time from the initiation of everolimus to disease progression or death, whichever occurred first.
Overall survival | Up to 24 months
  Defined from the initiation of everolimus to death of any cause.
Response rate | Up to 24 months
  Defined as the proportion of complete response and partial response per RECIST criteria.
Toxicity | Up to 24 months
  Any adverse events occurred during the treatment with study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Hee Ahn, MD, PhD, Principal Investigator — Asan Medical Center
Locations (8):
- South Korea (8):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Asan Medical Center, University of Ulsan College of Medicine, Seoul, N/A = Not Applicable
  - Yeongnam University College of Medicine, Daegu
  - Chungnam National University Hospital, Daejeon
  - Seoul National University Hospital, Seoul
  - Yonsei Cancer Center, Seoul
  - Korea University, Seoul
  - Samsung Medical Center, Seoul

REFERENCES:
- [Background] Edmonson JH, Ryan LM, Blum RH, Brooks JS, Shiraki M, Frytak S, Parkinson DR. Randomized comparison of doxorubicin alone versus ifosfamide plus doxorubicin or mitomycin, doxorubicin, and cisplatin against advanced soft tissue sarcomas. J Clin Oncol. 1993 Jul;11(7):1269-75. doi: 10.1200/JCO.1993.11.7.1269. PMID 8315424
- [Background] Verweij J, Lee SM, Ruka W, Buesa J, Coleman R, van Hoessel R, Seynaeve C, di Paola ED, van Glabbeke M, Tonelli D, Judson IR. Randomized phase II study of docetaxel versus doxorubicin in first- and second-line chemotherapy for locally advanced or metastatic soft tissue sarcomas in adults: a study of the european organization for research and treatment of cancer soft tissue and bone sarcoma group. J Clin Oncol. 2000 May;18(10):2081-6. doi: 10.1200/JCO.2000.18.10.2081. PMID 10811673
- [Background] Hartmann JT, Patel S. Recent developments in salvage chemotherapy for patients with metastatic soft tissue sarcoma. Drugs. 2005;65(2):167-78. doi: 10.2165/00003495-200565020-00002. PMID 15631540
- [Background] Santoro A, Tursz T, Mouridsen H, Verweij J, Steward W, Somers R, Buesa J, Casali P, Spooner D, Rankin E, et al. Doxorubicin versus CYVADIC versus doxorubicin plus ifosfamide in first-line treatment of advanced soft tissue sarcomas: a randomized study of the European Organization for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group. J Clin Oncol. 1995 Jul;13(7):1537-45. doi: 10.1200/JCO.1995.13.7.1537. PMID 7602342
- [Background] Le Cesne A, Judson I, Crowther D, Rodenhuis S, Keizer HJ, Van Hoesel Q, Blay JY, Frisch J, Van Glabbeke M, Hermans C, Van Oosterom A, Tursz T, Verweij J. Randomized phase III study comparing conventional-dose doxorubicin plus ifosfamide versus high-dose doxorubicin plus ifosfamide plus recombinant human granulocyte-macrophage colony-stimulating factor in advanced soft tissue sarcomas: A trial of the European Organization for Research and Treatment of Cancer/Soft Tissue and Bone Sarcoma Group. J Clin Oncol. 2000 Jul;18(14):2676-84. doi: 10.1200/JCO.2000.18.14.2676. PMID 10894866
- [Background] van Oosterom AT, Mouridsen HT, Nielsen OS, Dombernowsky P, Krzemieniecki K, Judson I, Svancarova L, Spooner D, Hermans C, Van Glabbeke M, Verweij J; EORTC Soft Tissue and Bone Sarcoma Group. Results of randomised studies of the EORTC Soft Tissue and Bone Sarcoma Group (STBSG) with two different ifosfamide regimens in first- and second-line chemotherapy in advanced soft tissue sarcoma patients. Eur J Cancer. 2002 Dec;38(18):2397-406. doi: 10.1016/s0959-8049(02)00491-4. PMID 12460784
- [Background] Clark MA, Fisher C, Judson I, Thomas JM. Soft-tissue sarcomas in adults. N Engl J Med. 2005 Aug 18;353(7):701-11. doi: 10.1056/NEJMra041866. No abstract available. PMID 16107623
- [Background] Wan X, Helman LJ. The biology behind mTOR inhibition in sarcoma. Oncologist. 2007 Aug;12(8):1007-18. doi: 10.1634/theoncologist.12-8-1007. PMID 17766661
- [Background] Motzer RJ, Escudier B, Oudard S, Hutson TE, Porta C, Bracarda S, Grunwald V, Thompson JA, Figlin RA, Hollaender N, Urbanowitz G, Berg WJ, Kay A, Lebwohl D, Ravaud A; RECORD-1 Study Group. Efficacy of everolimus in advanced renal cell carcinoma: a double-blind, randomised, placebo-controlled phase III trial. Lancet. 2008 Aug 9;372(9637):449-56. doi: 10.1016/S0140-6736(08)61039-9. Epub 2008 Jul 22. PMID 18653228
- [Derived] Yoo C, Lee J, Rha SY, Park KH, Kim TM, Kim YJ, Lee HJ, Lee KH, Ahn JH. Multicenter phase II study of everolimus in patients with metastatic or recurrent bone and soft-tissue sarcomas after failure of anthracycline and ifosfamide. Invest New Drugs. 2013 Dec;31(6):1602-8. doi: 10.1007/s10637-013-0028-7. Epub 2013 Sep 14. PMID 24037083